CLINICAL TRIAL: NCT02001532
Title: Arterial Stiffness and Complication Risk in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: 1-10-72-349-13
Record Dates: First submitted 2013-11-21; First posted 2013-12-05 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Complications; Diabetic Angiopathies; Diabetic Nephropathies
Keywords: Diabetes Mellitus, Type 2; Diabetes Complications; Diabetic Angiopathies; Diabetic Nephropathies; Myocardial Infarction; Stroke; Vascular Stiffness; Pulse Wave Analysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications; Diabetic Angiopathies; Diabetic Nephropathies; Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Whole blood Serum/plasma Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes type 2: Patients diagnosed with type 2 diabetes within 5 years from baseline (i.e. 10 years at follow-up)
- Healthy controls: Sex and age-matched healthy controls

SUMMARY:
Background

The prevalence and incidence of type 2 diabetes is increasing globally. A common complication of diabetes is the disease of the blood vessels, vascular diseases, which can cause disorders like myocardial infarction, stroke and kidney failure. Methods to detect early subclinical stages of macro-vascular disease are not yet available in a clinical setting.

Hypothesis

Arterial stiffness, an easy accessible vascular parameter, may provide additional prognostic information when evaluating risk profile for patients with diabetes type 2.

Aim

The aim of the project is to investigate the association between arterial stiffness and the occurrence and development of vascular complications in patients with type 2 diabetes. Specifically we want to investigate:

1. in a cross-sectional study, the association between arterial stiffness and subclinical atherosclerotic changes in the coronary arteries assessed by computed tomography (CT) and
2. in a longitudinal study, the predictive value of arterial stiffness on the development of subclinical cerebrovascular changes assessed by magnetic resonance imaging (MRI) and nephropathy assessed by urine analysis.

Methods

The study population consists of 100 patients with newly diagnosed type 2 diabetes and 100 age- and sex matched controls. The study participants were enrolled between 2008-2011 and extensively characterized i.a. with arterial stiffness (pulse wave velocity), MRI (white matter lesions and cerebral infarctions) and urine analysis (albuminuria). In this study we will enrol the same patients in a 5 year follow-up study in order to repeat above mentioned measurements. Furthermore, CT is used to investigate the coronary plaque burden of the participants (Agatston Score and Segment Involvement Score).

Results and Perspective

This project adds new insight into arterial stiffness as a predictor of the progression of micro- and macrovascular complications in patients with type 2 diabetes, and can potentially improve risk stratification and early strategies of intervention in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Diabetes, type 2, diagnosed within 5 years from baseline (cases)

Exclusion Criteria:

* Non-diagnosed diabetes (healthy controls)
* Acute or chronic infectious diseases
* Kidney failure (requiring dialysis)
* Pregnancy/breastfeeding
* Prior or concomitant cancer disease
* Contraindication for MRI (claustrophobia, magnetic implants or bodyweight above 120kg)
* Contraindication for CT (estimated glomerular filtration rate < 50 ml/min, Body Mass Index > 35 kg/m2, heart arrhythmia, heart failure, aorta stenosis, contraindications for beta blockage or nitroglycerin or failure to cooperate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients with type 2 diabetes (cases) were enrolled from the outpatient clinic of the Department of Endocrinology, Aarhus University Hospital between 2008-11.
  100 sex and age-matched healthy controls were recruited in the same time period through the local press.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
White matter lesions (MRI) | 5 years
  A surrogate marker of the risk of stroke
Albuminuria | 5 years
  A measure of kidney damage
Segment Involvement Score (CT) | Will be assessed within 3 weeks from enrollment
  Measure of coronary plaques and a surrogate marker of ischemic heart disease.
Agatston Score (CT) | Will be assessed within 3 weeks from enrollment
  Measure of calcium in the coronary arteries and a surrogate marker of ischemic heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Per L Poulsen, MD, Ph.D., dr.med.sci, Principal Investigator — Department of Medical Endocrinology, Aarhus University Hospital
Locations (1):
- Department of Medical Endocrinology, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Laugesen E, Rossen NB, Hoyem P, Christiansen JS, Knudsen ST, Hansen KW, Hansen TK, Poulsen PL. Reproducibility of pulse wave analysis and pulse wave velocity in patients with type 2 diabetes. Scand J Clin Lab Invest. 2013 Aug;73(5):428-35. doi: 10.3109/00365513.2013.800578. Epub 2013 Jun 18. PMID 23777282
- [Result] Laugesen E, Hoyem P, Stausbol-Gron B, Mikkelsen A, Thrysoe S, Erlandsen M, Christiansen JS, Knudsen ST, Hansen KW, Kim WY, Hansen TK, Poulsen PL. Carotid-femoral pulse wave velocity is associated with cerebral white matter lesions in type 2 diabetes. Diabetes Care. 2013 Mar;36(3):722-8. doi: 10.2337/dc12-0942. Epub 2012 Nov 5. PMID 23129135
- [Result] Laugesen E, Hoyem P, Christiansen JS, Knudsen ST, Hansen KW, Argraves WS, Hansen TK, Poulsen PL, Rasmussen LM. Plasma levels of the arterial wall protein fibulin-1 are associated with carotid-femoral pulse wave velocity: a cross-sectional study. Cardiovasc Diabetol. 2013 Jul 18;12:107. doi: 10.1186/1475-2840-12-107. PMID 23866070
- [Derived] Funck KL, Laugesen E, Ovrehus K, Jensen JM, Norgaard BL, Dey D, Hansen TK, Poulsen PL. Increased high-risk coronary plaque burden is associated with arterial stiffness in patients with type 2 diabetes without clinical signs of coronary artery disease: a computed tomography angiography study. J Hypertens. 2017 Jun;35(6):1235-1243. doi: 10.1097/HJH.0000000000001308. PMID 28441695